CLINICAL TRIAL: NCT02981420
Title: Implementing a Brief Suicide Intervention for High Risk Youth With Front-Line Juvenile Justice Staff
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rhode Island Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 927079; K23MH111606 (NIH)
Record Dates: First submitted 2016-11-28; First posted 2016-12-05 (Estimated); Last update posted 2017-03-06 (Actual); Status verified 2016-11

CONDITIONS: Suicide and Self Harm
MeSH Terms: conditions — Suicide; Self-Injurious Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Pre-intervention (No Intervention): Pre-intervention baseline comparison
- Safety Planning (Experimental): Intervention group
  Interventions: Behavioral: Safety planning
- Regression discontinuity (No Intervention): Subthreshold no intervention

INTERVENTIONS:
Behavioral: Safety planning — Safety Planning Intervention. This brief one-session intervention, based on cognitive behavioral principles, is designed to help individuals identify a concrete list of coping strategies and social supports that youth can utilize preceding or during a crisis to lower imminent risk of suicidal behavior. In youth who also report nonsuicidal self-injurious behavior (NSSI), the safety plan will address both suicidal and nonsuicidal behavior. The plan helps youth identify possible triggers to SI/crisis including self-monitoring of suicidal thoughts, feelings, and behaviors; advance planning to remove lethal means; determine distress tolerance/emotion regulation skills that may be helpful; identify accessible social supports to target hopelessness/sense of isolation; reinforce the commitment to seek treatment; and, how and where to access emergency care.
  Arms: Safety Planning

SUMMARY:
A youth's contact with the juvenile justice system represents an opportune moment for suicide screening and brief suicide intervention for indicated youth. This study will provide data on the novel implementation of an evidence-based brief suicide intervention, safety planning, administered by front-line juvenile court staff for suicidal court-involved non-incarcerated youth. Data will inform the dissemination and implementation of suicide brief interventions to be delivered by front-line staff at the time of mental health screening in the juvenile justice system. The proposed study is consistent with the NIMH Strategic Plan by testing an intervention for effectiveness in community settings (Strategy 3.3) and establishing a research-practice partnership to improve D&I of evidence-based MH services (4.2). The unique service delivery by JJ court staff also supports the NIMH goals to develop innovative service delivery models (Strategy 4.3) as well as validate a MH intervention for an underserved population (Strategy 4.1). This proposal also addresses the Healthy People 2020 goals of reducing suicide attempts (MHMD-2).

DETAILED DESCRIPTION:
Suicide and suicidal behaviors among youth in the United States represents a significant public health problem. Youth involved in the juvenile justice system have a greater burden of risk factors associated with suicide ideation and behaviors as compared to their non-justice involved peers, placing these youth at greater risk for suicide. Thus, the overall goal of this Mentored Patient-Oriented Research Career Development Award (K23) is to support the applicant in developing the skills to launch an independent research program focused on the dissemination and implementation of evidence-based interventions for court-involved non-incarcerated (CINI) youth involved in the juvenile justice system to reduce psychiatric morbidity. Specific training goals are: (1) engage in intensive clinical and research training to increase my expertise in conducting brief interventions for adolescent suicide, (2) develop expertise in dissemination and implementation strategies and research in the juvenile justice system, (3) achieve skills in mixed-method research methodology including design and analysis of studies to support causal inference when randomization is not possible. The applicant will pursue these goals through a combination of mentoring, didactics, and practical experience. Specific training goals for this 5-year-period will be achieved under the mentorship of Drs. Anthony Spirito (Brown University), Marina Tolou-Shams (UCSF), Gina Vincent (UMASS Medical School), and Peter Friedmann (Baystate Health). The objective of the proposed research study is to 1) identify individual-, administrative-, and system-level factors that promote or hinder uptake of a brief suicide intervention conducted by front-line juvenile justice staff with CINI youth and 2) implement an evidence-based brief intervention, safety planning, for suicidal CINI youth and evaluate its utility with these youth. In the Treatment Adaptation phase, 12 juvenile justice stakeholders will be interviewed pre- and post-intervention implementation, as well as 24 youth and 24 caregivers 3-months post-intervention, about the acceptability of the brief intervention in the juvenile court setting. In the Treatment Trial phase, we will examine the effectiveness of a safety planning intervention for indicated suicidal youth in reducing suicidal ideation, in reducing suicidal events (suicide attempts as well as emergency evaluations and psychiatric hospitalizations for suicidality), increased engagement in outpatient mental health treatment, and improved youth motivation for treatment. CINI juveniles, ages 12-17, (N=100 for baseline (historical control) cohort; N=100 for efficacy trial; N=100 for alternative causal design) and a caregiver will be recruited from the juvenile court to participate in the current study. CINI juveniles in the efficacy trial will receive the evidenced-based brief suicide intervention as part of standard of care and will be compared to historical control and alternative causal design. Baseline data will be collected as part of routine care. Youth and a caregiver will be re-assessed at 3 months subsequent to the juvenile's initial court appointment.

ELIGIBILITY:
Inclusion Criteria:

* Court-involved non-incarcerated (CINI) youth,
* ages 12-17
* Legal guardian available to consent for juvenile's participation,
* Juvenile is English speaking, and
* Juvenile flags in the caution or warning range of the MAYSI-2.

Inclusion for second cohort:

* Court-involved non-incarcerated (CINI) youth,
* ages 12-17
* Legal guardian available to consent for juvenile's participation,
* Juvenile is English speaking, and
* Juvenile does not flag in the caution or warning range of the MAYSI-2

Exclusion Criteria:

* observable cognitive, developmental delays, or psychosis that would interfere with completing consent, assessment or intervention, and
* Juvenile meets hospital level of care for imminent suicide risk.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2016-12; Primary Completion 2019-05 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Self-Injurious Thoughts and Behaviors Interview 2.0 (SITBI 2.0) Short Form | 3 months
  Structured interview designed to assess the presence, frequency, and characteristics of a broad array of self-injurious thoughts and behaviors
Suicide Ideation Questionnaire (SIQ) - Junior | 3 months
  assesses the frequency of suicidal ideation
Child and Adolescent Services Assessment | 3 months
  parent report of utilization of MH services and operationalized as a composite score of suicide attempts and emergency interventions for acute suicidality assessed by the Child and Adolescent Services Assessment (CASA)
Treatment Attendance | 3 months
  Attendance at first treatment appointment and total number of treatment sessions attended will be collected by contacting each juveniles' treatment provider at the 3-month follow-up
Recidivism | 3 months
  Collateral data gathered from court database). Juveniles' recidivism rates (e.g., new arrests), description of related charges (e.g., substance-related, property) and time detained/incarcerated

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Kemp, Ph.D., Principal Investigator — RIH/Brown University
Locations (1):
- Rhode Island Family Court, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No